CLINICAL TRIAL: NCT07173517
Title: Cost Profile and Budget Implications of Rechargeable Versus Non-rechargeable Sacral Neuromodulation Devices for Neurogenic Lower Urinary Tract Dysfunction
Acronym: SNM、NLUTD
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Aerospace Center Hospital (Other); Shandong Provincial Hospital (Other Government); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Beijing Hospital (Other Government); Xi'an Honghui Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Second Hospital of Jilin University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202505-101
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-07

CONDITIONS: Rechargeable Sacral Neuromodulation Device; Neurogenic Lower Urinary Tract Dysfunction
Keywords: neurogenic lower urinary tract dysfunction; cost-savings; sacral neuromodulation; rechargeable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No biological samples were involved and only patient information was collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- rechargeable group
- non-rechargeable group

SUMMARY:
Traditional sacral neuromodulation devices are not rechargeable. In recent years, new rechargeable sacral neuromodulation devices have been developed and put into the market. The aim of this study was to evaluate the cost savings of a rechargeable sacral neuromodulation device versus a non-rechargeable sacral neuromodulation device for the treatment of neurogenic lower urinary tract dysfunction.

DETAILED DESCRIPTION:
From August 2020 to January 2025, 41 rechargeable and 227 non-rechargeable SNM patients with neurogenic lower urinary tract dysfunction in ten centers were enrolled in this study. Demographic data, SNM treatment-related costs, and adverse events (e.g., treatment discontinuation, infection, surgical site pain, and lead dislocation or fracture) were recorded for each patient to estimate the costs of long-term SNM treatment with rechargeable versus nonrechargeable devices.

SPSS 25.0 software was used for statistical analysis of the data. Measurement data were expressed as mean ± SD, count data were expressed as cases (%), and paired t test was used for comparison before and after treatment in the group. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients with neurogenic lower urinary tract dysfunction who had failed conventional treatment
* obstructive urinary retention and contraindications to SNM

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: They were treated with rechargeable or non-rechargeable sacral neuromodulation devices
Sampling Method: Non-Probability Sample
Enrollment: 268 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Costs associated with sacral neuromodulation therapy | From August 2020 to January 2025
  Costs associated with sacral neuromodulation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided